CLINICAL TRIAL: NCT07235020
Title: A Multi-part, Multi-center PLATform Study to Assess the Efficacy, Safety, Tolerability and Pharmacokinetics of Anti-malarial Agents Administered as Monotherapy and/or Combination Therapy IN Participants With Uncomplicated Plasmodium Falciparum Malaria
Brief Title: Platform Study to Evaluate the Efficacy and Safety of Anti-malarial Agents in Participants With Uncomplicated Plasmodium Falciparum Malaria
Acronym: PLATINUM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CADPT13A12201_A1
Record Dates: First submitted 2025-11-14; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-10

CONDITIONS: Uncomplicated Plasmodium Falciparum Malaria
Keywords: single dose cure malaria; uncomplicated malaria; Plasmodium falciparum; platform study; PLATINUM
MeSH Terms: conditions — Malaria, Falciparum | interventions — INE963

STUDY DESIGN:
Masking Description: This study is open-label study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cohort A1: INE963 Dose Level 1 (Experimental): Cohort A1: INE963 Dose Level 1
  Interventions: Drug: INE963
- Cohort A1: INE963 Dose Level 2 (Experimental): Cohort A1: INE963 Dose Level 2
  Interventions: Drug: INE963
- Cohort A1: INE963 Dose Level 3 (Experimental): Cohort A1: INE963 Dose Level 3
  Interventions: Drug: INE963
- Cohort A1: INE963 Dose Level 4 (Experimental): Cohort A1: INE963 Dose Level 4
  Interventions: Drug: INE963

INTERVENTIONS:
Drug: INE963 — Administered via oral INE963

SUMMARY:
This is Cohort A1 of the Platform study (NCT05750628) to evaluate the efficacy and safety of INE963 in participants with uncomplicated Plasmodium falciparum malaria.

DETAILED DESCRIPTION:
The Cohort A1 of this Platfom study (NCT05750628) is an open-label, randomized, multi-arm monotherapy part evaluating a single oral administration of an anti-malarial agent (INE963) at 3 parallel dose levels followed by optional adaptive sequential dose level(s).

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients ≥18 years of age at screening.
2. Patients must have acute uncomplicated P. falciparum malaria mono infection at screening confirmed by a parasite count between 5,000 to 150,000 asexual parasite count/μl of blood for P. falciparum
3. Patients must weigh between 40 kg and 90 kg.
4. Axillary temperature ≥ 37.5ºC or oral/tympanic/rectal temperature ≥ 38.0ºC; or history of fever during the previous 24 hours.

Exclusion Criteria:

1. Patients with signs and symptoms of severe/complicated malaria at screening or mixed Plasmodium infection (i.e., infection with more than one malaria species) at screening
2. Moderate to severe anemia, chronic hemoglobinopathy (Hemoglobin level < 8 g/dL), or known chronic underlying disease such as sickle cell disease at screening
3. Known clinically significant liver disease (e.g., chronic hepatitis, liver cirrhosis (compensated or decompensated), history of hepatitis B or C, hepatitis A or B vaccination in the last 3 months, known gallbladder or bile duct disease, acute or chronic pancreatitis. Clinical or laboratory evidence of any of the following at screening:

   * AST/ALT > 3 x the upper limit of normal range (ULN), regardless of the level of total bilirubin
   * AST/ALT > 1.5 and ≤ 2 x ULN and total bilirubin is > ULN
   * Total bilirubin > 2 x ULN, regardless of the level of AST/ALT
4. Any known/suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection at screening.
5. Pregnant or nursing (lactating) women, women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using methods of effective contraception, and sexually active patients not willing to practice effective contraception.
6. History or current diagnosis of ECG abnormalities indicating significant risk of safety for patients participating in the study such as:

   * Concomitant clinically significant cardiac arrhythmias, e.g., sustained ventricular tachycardia, and clinically significant second or third degree AV block without a pacemaker
   * History of familial long QT syndrome or known family history of Torsades de Pointe.
   * Resting heart rate (physical exam or 12 lead ECG) < 50 bpm

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2024-01-23 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-02-21 (Actual)

PRIMARY OUTCOMES:
Parasite clearance time (PCT) | up to Day 7
  To assess the parasite clearance time (PCT) of oral doses of an anti-malarial agent administered as monotherapy in participants with uncomplicated P. falciparum malaria. PCT is defined as the time from the first positive blood slide at inclusion to the time of the first negative slide followed by two consecutive slides.

SECONDARY OUTCOMES:
PCR-corrected and uncorrected ACPR | Day 29
  To assess the 28-day cure rate of an anti malarial agent administered orally as monotherapy in participants with uncomplicated P. falciparum malaria.
Area under the concentration-time curve from time zero to the last measurable concentration sampling time (AUClast) | Day 22
  To characterize the pharmacokinetics (PK) of the anti-malarial agent administered orally as monotherapy.
Area under the concentration-time curve from time zero to infinity (AUCinf) | Day 22
  To characterize PK of the anti-malarial agent administered orally as monotherapy.
Maximum observed concentration (Cmax) | Day 22
  To characterize PK of the anti-malarial agent administered orally as monotherapy.
Time to reach maximum observed concentration (Tmax) | Day 22
  To characterize PK of the anti-malarial agent administered orally as monotherapy.
Elimination half-life (T1/2) | Day 22
  To characterize PK of the anti-malarial agent administered orally as monotherapy.
Total body clearance (CL/F) | Day 22
  To characterize PK of the anti-malarial agent administered orally as monotherapy.
Apparent volume of distribution (V/F) | Day 22
  To characterize PK of the anti-malarial agent administered orally as monotherapy.
Area under the concentration-time curve (AUC0-t) | Day 22
  To characterize PK of the anti-malarial agent administered orally as monotherapy.

CONTACTS AND LOCATIONS:
Locations (6):
- Novartis Investigative Site, Banfora, Burkina Faso
- Novartis Investigative Site, Azaguié, Côte d’Ivoire
- Novartis Investigative Site, Lambaréné, Gabon
- Novartis Investigative Site, Navrongo, Ghana
- Novartis Investigative Site, Kisumu, Kenya
- Novartis Investigative Site, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.